CLINICAL TRIAL: NCT02315781
Title: Parkinson's Disease Depression and tDCS
Brief Title: tDCS in Parkinson's Disease With Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources to conduct study withdrawn
Sponsor: Pacific Parkinson's Research Centre (Other)
Responsible Party: Principal Investigator, A. Jon Stoessl, Co-Director of the Centre for Brain Health UBC, Pacific Parkinson's Research Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H14-00867
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Depression; Parkinson's
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Active Comparator): active tDCS will be used on half of the study participants
  Interventions: Device: active tDCS
- Sham tDCS (Sham Comparator): Sham tDCS will be used on half of the study participants
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: active tDCS — transcranial direct current stimulation (tDCS), is a type of electrical stimulation for the brain
  Arms: Active tDCS
Device: Sham tDCS — Sham tDCS will appear exactly the same as active tDCS, but no stimulation will be administered.
  Arms: Sham tDCS

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disease that has effects on both movement and mental health. One of the most common mental health complications of PD is depression. Up to 30% of Parkinson's patients will experience depression at some point. We aim to investigate whether transcranial direct current stimulation (tDCS), a type of electrical stimulation for the brain, can improve depression in PD as well as improve motor function in PD.

DETAILED DESCRIPTION:
The purpose of this double-blind, randomized control design study is to investigate the efficacy of 15-sessions of tDCS (versus 15-sessions of sham tDCS) to treat depression in PD. We will also assess dopamine function in a smaller cohort of participants before and after their 15 sessions of tDCS by using PET scanning.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients,
2. are voluntary and competent to consent to treatment,
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of major depressive disorder (MDD),
4. have a diagnosis of PD according to the UK PD brain bank criteria,
5. are 19 years of age or more,
6. have a score > 13 on the Beck Depression Inventory-II (BDI-II),
7. still have depressive symptoms after 6 weeks or more of antidepressant (SSRI) medication treatment (and on a stabilized dose of at least 4 weeks),
8. are able to adhere to the treatment schedule,
9. are proficient in written and verbal English.

Exclusion Criteria:

1. have a history of substance dependence or abuse within the last 6 months,
2. have a concomitant significant unstable medical illness,
3. have active suicidal intent,
4. have any history of seizure or medication-resistant epilepsy in the family,
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD,
7. have failed a course of ECT in the current episode or previous episode,
8. have received tDCS or other neurostimulation therapy for any previous indication due to the potential compromise of expectancy effects,
9. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes, or developmental disorder,
10. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed,
11. are taking a non-SSRI antidepressant medication,
12. are pregnant (women of childbearing age only).

Exclusion Criteria for PET:

1. unable to tolerate staying off anti-parkinsonian medication for 12-18 hours pre-PET scan,
2. have a history of radiation therapy treatment or other high amounts of radiation.

Exclusion Criteria for MRI:

* Artificial heart valve;
* Brain aneurysm clip;
* Electrical stimulator for nerves or bones;
* Ear or eye implant;
* Implanted drug infusion pump;
* Coil, catheter, or filter in any blood vessel;
* Orthopedic hardware (artificial joint, plate, screws);
* Other metallic prostheses;
* Shrapnel, bullets, or other metal fragments;
* Surgery or tattoos (including tattooed eyeliner) in the last six weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
HAMD score | 12 weeks
  an assessment of the severity of depression

SECONDARY OUTCOMES:
Dopamine levels | 12 weeks
  PET scanning will be used to assess dopamine levels before and after sham/active tDCS in 20 participants

CONTACTS AND LOCATIONS:
Overall Officials: A.J Stoessl, MD, Principal Investigator — Pacific Parkinson's Research Centre
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada